CLINICAL TRIAL: NCT01900249
Title: A Phase 2, Multi-Center, Randomized, Double-Masked, Placebo-Controlled Clinical Study to Assess the Safety and Efficacy of 0.2% and 0.5% R932348 Ophthalmic Solutions in Patients With Keratoconjunctivitis Sicca
Brief Title: To Assess the Safety and Efficacy of R932348 Ophthalmic Solutions in Patients With Keratoconjunctivitis Sicca
Acronym: DROPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-932348-003
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Keratoconjunctivitis Sicca
MeSH Terms: conditions — Keratoconjunctivitis Sicca

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- R348 Ophthalmic Solution, 0.2% (Active Comparator): R348 Ophthalmic Solution, 0.2%
  Interventions: Drug: R348 Ophthalmic Solution, 0.2%
- R348 Ophthalmic Solution, 0.5% (Active Comparator): R348 Ophthalmic Solution, 0.5%
  Interventions: Drug: R348 Ophthalmic Solution, 0.5%
- Placebo (Placebo Comparator): Placebo Ophthalmic Solution, 1 drop per eye twice a day for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: R348 Ophthalmic Solution, 0.2% — R348 Ophthalmic Solution, 0.2% 1 drop per eye twice a day for 12 weeks.
  Other Names: R932348
  Arms: R348 Ophthalmic Solution, 0.2%
Drug: R348 Ophthalmic Solution, 0.5% — R348 Ophthalmic Solution, 0.5% 1 drop per eye twice a day for 12 weeks.
  Other Names: R932348
  Arms: R348 Ophthalmic Solution, 0.5%
Drug: Placebo — Placebo Ophthalmic Solution 1 drop per eye twice a day for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether 0.2% and 0.5% R348 Ophthalmic Solutions are safe and effective in the treatment of Patients with Keratoconjunctivitis Sicca.

ELIGIBILITY:
Inclusion Criteria:

* A history of dry eye (based on the date of initial dry eye symptoms)
* Use of over-the-counter (OTC) and/or prescription eye drops for dry eye symptoms
* Corneal fluorescein staining score of at least 2 in the inferior region

Exclusion Criteria:

* History of, or a concurrent clinically significant illness, medical condition (other than Keratoconjunctivitis Sicca or Sjögren's syndrome), or laboratory abnormality that, in the Investigator's opinion, could affect the conduct of the study.
* Use of ophthalmic cyclosporine within 45 days of Visit 1.
* Use of any topical ophthalmic steroid within 2 weeks of Visit 1.
* Have worn contact lenses or anticipate using contact lenses during the study.
* Have a condition or be in a situation that the Investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.
* Have a history of alcohol or substance abuse that, in the judgment of the Investigator, may impair or risk the subject's full participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Magilavy, MD, Study Director — Rigel Pharmaceuticals,Inc.
Locations (20):
- United States (20):
  - Sall Research Medical Center, Artesia, California
  - North Bay Eye, Petaluma, California
  - Martel Medical Eye Group, Rancho Cardova, California
  - Specialty Eye Care, Parker, Colorado
  - International Research Center, Brandon, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Clayton Eye Center, Morrow, Georgia
  - Coastal Research Associates, Roswell, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Chicago Cornea Consultants, Hoffman Estates, Illinois
  - Koffler Vision Group, Lebanon, Kentucky
  - Taustine Eye Center, Louisville, Kentucky
  - Comprehensive Eye Care, Ltd/Vision Research Institute, LLC, Washington, Missouri
  - Mundorf Eye Center, Charlotte, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates, PA, Charlotte, North Carolina
  - Cornerstone Eyecare, High Point, North Carolina
  - Abrams Eye Center, Cleveland, Ohio
  - Glaucoma Consultants and Center for Eye Research, Mt. Pleasant, South Carolina
  - Chattanooga Eye Institute, Chattanooga, Tennessee
  - Eye Clinics of South Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | R348 Ophthalmic Solution, 0.2% | R348 Ophthalmic Solution, 0.5% | Placebo
Started | 67 | 68 | 69
Completed | 64 | 63 | 65
Not Completed | 3 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | R348 Ophthalmic Solution, 0.2% | R348 Ophthalmic Solution, 0.5% | Placebo | Total
Number analyzed (Participants) | 67 | 68 | 69 | 204
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (11.59) | 63.3 (11.5) | 61.5 (15.2) | 62.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 54 | 162
  Male | 13 | 14 | 15 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change of Corneal Fluorescein Staining of the Inferior Cornea Region.
Description: Change from baseline (Visit 3) of inferior region CFS score at 12 weeks. Inferior region CFS score range 0-4, where '0' represents no fluorescein staining and '4' represents severe staining on the cornea.
Time Frame: Baseline to Week 12
Population: The intent to treat population (ITT) included all randomized subjects who administered study medication. The primary analysis was performed on the ITT population.
Measure: Mean (95% Confidence Interval); unit: units on a scale (Likert)
Arm/Group | R348 Ophthalmic Solution, 0.2% | R348 Ophthalmic Solution, 0.5% | Placebo
Number analyzed (Participants) | 67 | 68 | 69
units on a scale (Likert) | -1.00 [-3.0 to 1.0] | -0.78 [-2.5 to 1.0] | -0.78 [-2.5 to 1.0]

ADVERSE EVENTS:
Time Frame: The AE reporting period begins with the first dose of double blind study drug and ends with the final study (Day 91) visit.
Arm/Group | R348 Ophthalmic Solution, 0.2% | R348 Ophthalmic Solution, 0.5% | Placebo
Serious Adverse Events (participants affected / at risk) | 3/67 | 1/68 | 2/69
Other Adverse Events (participants affected / at risk) | 36/67 | 46/68 | 31/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R348 Ophthalmic Solution, 0.2% (N=67) | R348 Ophthalmic Solution, 0.5% (N=68) | Placebo (N=69)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Malignant hyperthermia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R348 Ophthalmic Solution, 0.2% (N=67) | R348 Ophthalmic Solution, 0.5% (N=68) | Placebo (N=69)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye Discharge (Eye disorders) | 3 (3) | 3 (3) | 2 (2)
Conjunctival Hyperaemia (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Meibomianitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Periorbital Oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 3 (3) | 0 (0) | 1 (1)
Conjunctival Cyst (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctival Disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis Allergic (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye Pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Punctate Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Trichiasis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 2 (3)
Corneal Abrasion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Salivary Duct Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Instillation Site Pain (General disorders) | 17 (20) | 35 (37) | 3 (3)
Instillation Site Pruritus (General disorders) | 1 (1) | 4 (4) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
instillation Site Paraesthesia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Instillation Site Discomfort (General disorders) | 4 (5) | 0 (0) | 2 (2)
Hyperthermia Malignant (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Track Infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis Bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post Procedural Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Urine Analysis Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Intraocular Pressure Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Manifest Refraction (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral Disc Protusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Viith Nerve Paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tooth Extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Rotator Cuff Repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less